CLINICAL TRIAL: NCT02846909
Title: The Effect of Adjunctive Use of Vaginal Progesterone After Cerclage on Prevention of 2nd Trimester Miscarriage
Brief Title: The Vaginal Progesterone and Cerclage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCR
Record Dates: First submitted 2016-07-23; First posted 2016-07-27 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Abortion
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal progesterone group (Active Comparator): Will receive progesterone pessaries 400 mg once daily vaginally
  Interventions: Drug: Progesterone
- No progesterone group (No Intervention): Will receive nothing

INTERVENTIONS:
Drug: Progesterone — 400mg progesterone pessaries
  Arms: Vaginal progesterone group

SUMMARY:
Pregnancy loss in the second trimester is not uncommon. About 2-3% of pregnancies will be lost in the second trimester, which is much lower than in the first trimester. Once a pregnancy reaches 20 weeks gestation, less than 0.5% will end in a fetal demise.

Congenital fetal abnormalities and maternal anatomic factors as immunologic factors, infection, and thrombophilia should be considered; however, a reason and its result connection may be difficult to be established.

Cervical incompetence means that the cervix is weak and unable to remain closed during the pregnancy. While cerclage may provide a degree of support to a 'weak' cervix, its role in maintaining the cervical length and the endocervical mucus plug as a mechanical barrier to ascending infection may be more important.

Cervical cerclage is performed usually in women with a history of mid-trimester abortion or spontaneous preterm birth due to cervical 'incompetence', with the aim of preventing recurrent loss.

Cerclage is a commonly performed as a prophylactic intervention used by most obstetricians despite the absence of a well-defined population for whom there is clear evidence of benefit. Furthermore, there is little consensus on the optimal cerclage technique and timing and type of suture placement.

The Progesterone is known to have an inhibitory action on uterine contractility and is thought to play a main role in the maintenance of pregnancy until term. Progesterone is also able to modify the ultrastructural organisation of the myometrium by inhibiting the gap junctions, and preventing muscular contraction.

Different routes of administration of progesterone have been described in the literature. These include weekly intramuscular injections from 16 to 20 weeks through to 36 weeks and daily vaginal progesterone suppositories from 24 weeks to 34 weeks of gestation.

A recently published Cochrane review further confirmed the beneficial effects of progesterone in infant health following administration in women considered to be at increased risk of preterm birth due either to past history of preterm birth or when a short cervix was identified on ultrasound.

However; most of these published studies have been conducted to test the effect of progestational agents for the prevention of preterm labor not miscarriage.

Doppler ultrasonography is use to evaluate blood flow. In the field of perinatology, Doppler ultrasonography has been used to assess fetal well-being, especially in intra-uterine growth retardation and fetal anemia, and it plays an important role in managing of these conditions

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 - 35 years old.
* Pregnant from (12- 14 weeks) gestation.
* Singleton pregnancy.
* The pregnant women who have a history of second trimester pregnancy loss with painless cervical dilatation or have prior cerclage placement for cervical insufficiency or have a history of spontaneous preterm.

Exclusion Criteria:

* Multiple gestations.
* Congenital fetal malformation in the current pregnancy.
* Women with history of thromboembolism or bleeding disorders.
* Uncontrolled diabetes mellitus.
* Chromosomal abnormalities affecting one of the couples.
* Women refuse to participate in the study
* Antiphospholipid syndrome

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
The frequency of spontaneous abortion before 28 weeks | 14 weeks
  number of women aborted before 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Eleje GU, Eke AC, Ikechebelu JI, Ezebialu IU, Okam PC, Ilika CP. Cervical stitch (cerclage) in combination with other treatments for preventing spontaneous preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2020 Sep 24;9(9):CD012871. doi: 10.1002/14651858.CD012871.pub2. PMID 32970845
- [Derived] Ali MK, Ahmed SE, Sayed GH, Badran EY, Abbas AM. Effect of adjunctive vaginal progesterone after McDonald cerclage on the rate of second-trimester abortion in singleton pregnancy: a randomized controlled trial. Int J Gynaecol Obstet. 2020 Jun;149(3):370-376. doi: 10.1002/ijgo.13148. Epub 2020 Apr 29. PMID 32246762